CLINICAL TRIAL: NCT04265001
Title: Effectiveness of Topical Hyaluronic Acid Versus Chlorhexidine Mouthwashes in the Treatment of Recurrent Aphthous Stomatitis: A Randomized Clinical Trial
Brief Title: Topical Hyaluronic Acid and Recurrent Aphthous Stomatitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Zakaria Ibrahium Mohammed, Lecturer of Oral Medicine and Periodontology, Cairo University, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mai Zakaria Ibrahium
Record Dates: First submitted 2020-02-09; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Recurrent Aphthous Stomatitis
Keywords: recurrent aphthous stomatitis; chlorhexidine; hyaluronic acid; pain; topical
MeSH Terms: conditions — Stomatitis, Aphthous; Pain | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The clinical outcomes were assessed by an investigator masked about the treatment modality that has been used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Topical cholrhexidine hydrochloride 125 mg/100 ml available commercially (Hexitol; Arab Drug Company for Pharmaceutical and Chemical Industries, Cairo, Egypt) mouthwash. Topical cholrhexidine hydrochloride mouthwash treatment has been repeated three times per day for one week.
  Interventions: Drug: Hyaluronic acid in the form of hyaluronan sodium 25 mg/100 ml as a mouthwash
- Hyaluronic acid group (HA group) (Experimental): Topical hyaluronic acid in the form of hyaluronan sodium 25 mg/100 ml as a mouthwash (Aftamed; Bioplaxpharma, UK).Topical hyaluronic acid mouthwash treatment has been repeated three times per day for one week.
  Interventions: Drug: Hyaluronic acid in the form of hyaluronan sodium 25 mg/100 ml as a mouthwash

INTERVENTIONS:
Drug: Hyaluronic acid in the form of hyaluronan sodium 25 mg/100 ml as a mouthwash — Topical mouthwash used three times daily for one week and patients were not allowed to eat or drink for one hour after rinsing.
  Other Names: (Aftamed; Bioplaxpharma, UK)

SUMMARY:
This study was conducted to estimate the hypothesis that the topical hyaluronic acid mouthwash have no role in the treatment of recurrent aphthous stomatitis

DETAILED DESCRIPTION:
Recurrent aphthous stomatitis (RAS) is a common and widely recognized disorder involving the oral mucosa. It occurs typically as a single or multiple well-defined painful self-limiting ulcerative lesions influencing the nonkeratinized oral mucous membrane surrounded by red halo. The prevalence of RAS is up to 25% in the world population, with recurrence rate of 50% every 3 mouths. The exact cause of RAS is uncertain, and accordingly numerous components are as yet being implicated such as genetic, hormonal, traumatic, nutritional, allergic, immunological, and psychological factors.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were as follows:

* Age 18-30 years.
* Minimum of 2 years of RAS history, with active ulcer less than 48 hours of recurrent aphthous stomatitis.

Exclusion Criteria:

* known history of hypersensitivities to Chlorhexidine or hyaluronic acid.
* Use of any medication as a treatment for the present active ulcer.
* Smoking and presence of systemic diseases such as Behçet disease, anemia, Crohn's disease, ulcerative colitis, acquired immune deficiency syndrome, and liver or kidney disease.
* Pregnant or breast-feeding women.
* Stomach ulcer, duodenal ulcer, and inflammation of the stomach or the esophagus.
* Treatment with systemic nonsteroidal anti-inflammatory drugs, systemic steroids or other immune modulatory agents, oral antihistamines, or systemic antibiotics in the previous 3 months.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Pain score | one week
  Pain assessment scale, visual analog scale (VAS) comprising of a 10-cm straight line among ends, with 0 representing no pain (better outcome) and 10 for intolerable pain (worse outcome) after irritation of the ulcer with the periodontal probe.

SECONDARY OUTCOMES:
Ulcer size | one week
  The ulcer size was evaluated by determining the distance between two opposed boundaries of the ulcer edge, using a periodontal probe in millimeters.Score for clinical improvement of the sign where high values indicate worse outcome but low values indicate better outcome.
Duration of healing | one week
  period of the ulceration for complete healing

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Because the research not published yet.